CLINICAL TRIAL: NCT05198739
Title: Feasibility Study of the Pilot Implementation of the Video Interaction Project in Brazil
Brief Title: Video Interaction Project in Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-00057
Record Dates: First submitted 2021-12-10; First posted 2022-01-20 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Parenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video Interaction Project (VIP) Group (Experimental): Parent-Child dyads will participate in a Video Interaction Project to encourage parenting practices/relationships and child development by promoting positive parenting practices.
  Interventions: Other: Video Interaction Project (VIP) program

INTERVENTIONS:
Other: Video Interaction Project (VIP) program — Video Interaction Project (VIP) is a strengths-based, family-centered intervention designed to enhance parenting practices/relationships and child development by promoting positive parenting practices such as pretend play, shared reading, and daily routines. In VIP's core component, a VIP coach video-records the parent / child for 3-5 minutes playing/reading with a provided toy and/or book, then reviews the video with the parent to facilitate self-reflection on the interaction and identifies and reinforces strengths. In the US, VIP is delivered in the context of pediatric primary care visits, with a COVID-19 remote adaptation (see Section 6 for details). Research staff will delivery VIP through video calls with subjects in Brazil.

SUMMARY:
Early exposure to poverty is associated with adverse impacts on long-term educational achievement. Support of positive parenting is a key strategy to prevent emergence of socioeconomic disparities in child development. This study will assess the feasibility of the pilot implementation of an evidence-based parenting program designed to prevent disparities in child development, the Video Interaction Project (VIP), in Brazil, as an exemplar low- and middle-income country (LMIC), and explore changes in parenting and child outcomes after participation in the program.

DETAILED DESCRIPTION:
This international study will be conducted in Southern Brazil. After translation and cultural adaptation of VIP materials (Aim 1), a qualitative investigation of VIP implementation feasibility (Aim 2) will be conducted using semi-structured interviews and observation of engagement for approximately 50 caregiver-child dyads with children 0-5 years who will participate in 3 VIP sessions. To explore changes in parenting and child outcomes (Aim 3), dyads enrolled in the study (for Aim 2) will complete assessments pre- and post-participation in 3 VIP sessions.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver-child dyads with at least one child age 0 to 5 years;
* Caregiver can be contacted (has a working phone); and
* Caregiver is 18 years old or older.
* Child is 1 day to 5 years old

Exclusion Criteria:

* Caregiver is under 18 years old; and
* Child has a neurodevelopmental disability or known or suspected genetic syndrome

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Change in the Percentage of Acceptance of the Video Interaction Project | Baseline Visit, Visit 4 (7 months)
  Semi-structured interviews (approximately 40-60 min) conducted. Caregivers will share their opinions about activities, provided materials, barriers/facilitators to participation and use of intervention strategies in the home. Interviews will be audio recorded, transcribed, and translated from Brazilian Portuguese to English. Guides for the semi structured interviews have been developed based on previous studies and theoretical frameworks.
Change in Parenting practices in Cognitive stimulation | Baseline Visit, Visit 4 (7 months)
  StimQ - Infant survey will be used to evaluates reading, teaching, responsivity with the caregivers through a video call. The survey consist of 4 subscales, which are summed together for a total score (StimQ2-I range 0-42)
Changes in Parent-child interactions during reading | Baseline Visit, Visit 4 (7 months)
  Adult-Child Interactive Reading Inventory (ACIRI) assesses both adult and child behaviors in three categories that research has identified as critical: Enhancing Attention to Text, Promoting Interactive Reading and Supporting Comprehension, and Using Literacy Strategies. An observational measure where caregivers and children are observed and given an score (3 = most of the time, 2 =some of the time , 1 = infrequently, 0= not at all)
Change in Parent Reading Belief of their children | Baseline Visit, Visit 4 (7 months)
  The Parent Reading Belief Inventory (PRBI) is a self-reporting instrument that assess parents' beliefs about the frequency, quality, and importance of their child's literacy activities. The 42-item instrument provides seven subscales: positive affect, verbal participation, resources, teaching efficacy, knowledge base, environmental input, and reading instruction.

SECONDARY OUTCOMES:
Change in Depression in Caregivers | Baseline Visit, Visit 4 (7 months)
  The Edinburgh Postnatal Depression Scale (EPDS) is a questionnaire originally developed to assist in identifying possible symptoms of depression in the postnatal period.It is a 10-item questionnaire where women are asked to answer each question in terms of the past seven days. A score is calculated by adding the individual items for each question, the a score of 10 or above is commonly considered "possible depression."
Change in Stress in Caregivers | Baseline Visit, Visit 4 (7 months)
  The Perceived Stress Scale (PSS-10) is a 10-item questionnaire used to assess stress levels in young people and adults aged 12 and above. Respondents are asked how often they felt a certain way on a five-point scale from 'never' to 'very often'. (Never = 0, Almost never = 1, Sometimes = 2, Fairly often = 3, Very often = 4).The PSS score is then obtained by summing across all items. Higher scores indicate higher levels of perceived stress.
Child Development (CS) | Baseline Visit, Visit 4 (7 months)
  Development of the Dimensional Inventory of Child Development Assessment (IDADI) assess child development of children from zero to 72 months of age through parental reports covering Cognitive, Motor (Gross and Fine), Communication and Language (Receptive and Expressive), Socioemotional and Adaptive Behavior domains. A three-point Likert scale was established where: yes (2-points); sometimes (1-point) ; and no (0-point) to indicate if the skill was mastered.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Mendelsohn, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to Alan.Mendelsohn@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.